CLINICAL TRIAL: NCT00115232
Title: Inflammatory Profiles of Children at High Risk for Atherosclerosis
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Sandra A. Daugherty Foundation (Other)
Responsible Party: Sarah de Ferranti, MD MPH, Children's Hospital Boston
Other Study IDs: 04-03-044
Record Dates: First submitted 2005-06-21; First posted 2005-06-22 (Estimated); Last update posted 2008-01-16 (Estimated); Status verified 2008-01

CONDITIONS: Cardiovascular Disease; Metabolic Syndrome X; Hypercholesterolemia; Inflammation
Keywords: cardiovascular disease; metabolic syndrome; hypercholesterolemia; child; family history; inflammation
MeSH Terms: conditions — Cardiovascular Diseases; Metabolic Syndrome; Hypercholesterolemia; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fasting serum samples, frozen.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: Children without family history of early atherosclerosis
- 2: Children with family history of early atherosclerosis.
- 3: Parents of children without family history of early atherosclerosis
- 4: Parents of children with family history of early atherosclerosis

SUMMARY:
The purpose of this study is to evaluate levels of inflammatory mediators in children at risk for cardiovascular disease due to family history. We are measuring inflammatory markers in two groups of children and their parents: children with a family history of early atherosclerotic heart disease (cases), and healthy children without such a family history (controls). The design is a cross-sectional study, gathering a fasting blood sample and clinical and behavioral data on children and a parent.

DETAILED DESCRIPTION:
Family history is a well known risk factor for early atherosclerosis. Whether inflammation plays a role in the increased risk of family history is not known. In this prospective single-center study, we are recruiting children with and without a family history of premature atherosclerotic disease, defined as occurring < 55 years in males and <65 years in females. Children are recruited primarily from a pediatric preventive cardiology clinic at Children's Hospital Boston. We measure anthropomorphic characteristics, fasting lipid profiles and inflammatory marker levels, including high sensitivity C-reactive protein (hsCRP), intracellular adhesion molecule 1 (ICAM-1), P-selectin, and tumor necrosis factor alpha receptor 2 (TNFαR2).

In this sample of high-risk overweight children, Lp(a) and inflammatory markers could reflect cardiovascular risk outside lipid profiles.

ELIGIBILITY:
Inclusion Criteria:

* Age 8-21 years
* Parent able to participate
* Fasting state
* Live locally

Exclusion Criteria:

* Taking medication that may alter cholesterol levels or inflammatory state
* Past or present inflammatory illnesses

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Primarily children referred to preventive cardiology clinic.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2004-07; Primary Completion 2006-10 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah D. de Ferranti, MD MPH, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States